CLINICAL TRIAL: NCT03380585
Title: Postoperative Pain Assessment After Foraminal Enlargement Using Protaper Next and Reciproc File Systems.
Brief Title: Postoperative Pain and PTN and Reciproc
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Isparta Military Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IAH-4
Record Dates: First submitted 2017-12-15; First posted 2017-12-21 (Actual); Last update posted 2018-03-12 (Actual); Status verified 2017-12

CONDITIONS: Apical Periodontitis; Dental Pulp Necrosis
MeSH Terms: conditions — Periapical Periodontitis; Dental Pulp Necrosis

STUDY DESIGN:
Who Masked: Participant
Masking Description: Single-blinded (Participant)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reciproc (Experimental): Endodontic treatment will be performed in teeth with necrotic pulp and periapical periodontitis. Local anaesthesia will be provided (2% Novocaine with 1:80,000 epinephrine), isolation with rubber dam and standard access cavity preparation will be done.Using 2.5 % sodium hypochlorite, canal negotiation will be done. Coronal flaring with # 2 and #3 Gates-Glidden drills will be done. The canals will be obturated with gutta-percha and epoxy resin sealer. The treatments will be carried out in single-visit. In this group, intervention will be carried out by the Reciproc motor (VDW, Germany) and Reciproc single-file system. The intervention is foraminal enlargement with the Reciproc single-file system.
  Interventions: Procedure: Reciprocating single-file system
- ProTaper Next (Active Comparator): The active comparator is foraminal enlargement with the ProTaper Next multi-file system. Endodontic treatment is identical to experimental group except file systems used. In this group, ProTaper Next multi-file system will be used in enlarging apical foramina.
  Interventions: Procedure: Rotational multi-file system.

INTERVENTIONS:
Procedure: Reciprocating single-file system — After determining the working length, a flexible size 30 K-file will be inserted 1 mm beyond the WL and the apical foramen will be enlarged.The device in the experimental group moves in CW and CCW direction with different angles. It is a single-file endodontic file system. The intervention is reciprocating single-file system. A Reciproc single-file will be used for enlarging apical foramen. In the active comparator group, a continuous rotational multi-file system, ProTaper Next, will be used in enlarging apical foramen.
  Other Names: Reciproc
  Arms: Reciproc
Procedure: Rotational multi-file system. — After determining the working length, a flexible size 30 K-file will be inserted 1 mm beyond the WL and the apical foramen will be enlarged. In this group, a continuous rotational multi-file system, ProTaper Next, will be used in enlarging apical foramen.
  Other Names: ProTaper Next
  Arms: ProTaper Next

SUMMARY:
In this clinical trial, the researchers will investigate the effect of single-file reciprocating file system (Reciproc) versus multi-file rotational file systems (ProTaper Next) on the postoperative pain in adult patients who have necrotic pulp and apical periodontitis. The participants will be assigned by chance to separate groups that compare 2 different treatments, reciprocating single-file system (Reciproc) and rotational multi-file system (ProTaper Next).

DETAILED DESCRIPTION:
The infected root canal treatments will be performed using one-visit approach with either a reciprocating single-file system or a continuous rotational multi-file system. Foraminal enlargement will be perfomed using either Reciproc or ProTaper Next file systems. The root canals will be completed in single-visit. The patients will record their postoperative pain during the follow-up period using a VAS scale.

ELIGIBILITY:
Inclusion Criteria:

Participants who have in their mandibular or maxillary molar teeth necrotic pulp and apical periodontitis.

Exclusion Criteria:

Pregnancy, drug hypersensitivity, cardiac problems, previously performed endodontics treatment.

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-03-01 (Actual); Study Completion 2018-03-02 (Actual)

PRIMARY OUTCOMES:
4-step pain intensity measures using a Visual Analog Scale (VAS). | 7 days
  The severity of pain in 1-7 days according to the VAS: 0 no pain, 1-3 mild pain, 4-7 moderate pain, 7-10 severe pain.

SECONDARY OUTCOMES:
The number of patients taking an analgesic following the endodontics treatment. | 7 days
  The patients were asked to take an analgesic in the 7 days of time frame.

CONTACTS AND LOCATIONS:
Overall Officials: Ibrahim E YAYLALI, PhD, Study Director — Isparta Military Hospital
Locations (1):
- Isparta Military Hospital, Isparta, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes